CLINICAL TRIAL: NCT00732004
Title: Time Course Comparison of Contact Lens Maintenance Systems for Hydrogel Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Clinical Vision Research Australia (Other); Alcon Research (Industry)
Responsible Party: Carol Lakkis, Clinical Vision Research Australia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H08 002
Record Dates: First submitted 2008-08-08; First posted 2008-08-11 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- 1 (Experimental): Group 1
  Interventions: Device: Silicone Hydrogel Contact Lenses
- 2 (Experimental): Group 2
  Interventions: Device: 1x PMBH preserved MPS
- 3 (Experimental): Group 3
  Interventions: Device: 1x Polyquad/Aldox MPS

INTERVENTIONS:
Device: Silicone Hydrogel Contact Lenses
  Arms: 1
Device: 1x PMBH preserved MPS
  Arms: 2
Device: 1x Polyquad/Aldox MPS
  Arms: 3

SUMMARY:
The principal aim of this project is to determine the time course of development of contact lens and contact lens case contamination during daily wear of silicone hydrogel lenses. The secondary aim of the study is to determine whether the time course of development of contact lens and contact lens case contamination varies between two different contact lens care systems.

ELIGIBILITY:
Inclusion Criteria:

* Distance contact lens prescription between +8.00 and -10.00D.
* Cylindrical component of refractive error no greater than 1.25D in either eye.
* Vision correctable to 6/12 (0.30 logMAR) or better in each eye.
* Healthy normal eyes without anterior segment infection, inflammation or abnormality, or significant slitlamp findings.

Exclusion Criteria:

* Concurrent ocular medication
* Eye injury or surgery within twelve weeks immediately prior to enrolment.
* Current ocular irritation that would preclude contact lens fitting.
* Evidence of systemic or ocular abnormality, infection or disease likely to affect successful wear of contact lenses or use of their accessory solutions.
* Pregnant, lactating or planning a pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Vision Research Australia, Melbourne, Victoria, Australia